CLINICAL TRIAL: NCT05105243
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Single and Multiple Doses of CVN766 in Healthy Subjects
Brief Title: Phase 1 SAD/MAD Study of CVN766 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CVN-766
Record Dates: First submitted 2021-09-29; First posted 2021-11-03 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Safety Issues; Tolerance
Keywords: PK; Efficacy

STUDY DESIGN:
Intervention Model Description: For the single-dose regimen, approximately 40 healthy male or female participants will be enrolled in 1 of 5 single-dose cohorts (designated as S1 through S5, respectively) in an ascending fashion. Each cohort will consist of 8 participants randomized to CVN766 or placebo, whereby 6 participants will receive a single oral dose of CVN766 suspension, and 2 participants will receive a matching placebo suspension under overnight fasted conditions.
  For the multiple-dose regimen, approximately 24 healthy male and female participants age 18 to 50 years old will be enrolled in 1 of the 3 multiple-dose cohorts (designated as M1 through M3, respectively) in an ascending fashion. The dose levels planned to be studied in the multiple-dose regimen are 45, 125, and 250 mg CVN766 for multiple-dose cohorts M1 through M3, respectively.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind. placebo-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Cohort 1 (Active Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 5 mg.
  Interventions: Drug: CVN766
- SAD Cohort 2 (Active Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 15 mg.
  Interventions: Drug: CVN766
- SAD Cohort 3 (Active Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 45 mg.
  Interventions: Drug: CVN766
- SAD Cohort 4 (Active Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 125 mg.
  Interventions: Drug: CVN766
- SAD Cohort 5 (Placebo Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 250 mg.
  Interventions: Drug: CVN766
- MAD Cohort 1 (Active Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 45mg.
  Interventions: Drug: CVN766
- MAD Cohort 2 (Placebo Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 125 mg.
  Interventions: Drug: CVN766
- MAD Cohort 3 (Placebo Comparator): Each dose cohort: 8 participants (6 active:2 placebo). 250 mg.
  Interventions: Drug: CVN766

INTERVENTIONS:
Drug: CVN766 — highly selective orexin-1 receptor (Ox1R) antagonist

SUMMARY:
Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Single and Multiple Doses of CVN766 in Healthy participants.

DETAILED DESCRIPTION:
Study Design:

This is a Phase 1, randomized, double-blind, placebo-controlled, single- and multiple-dose ascending study in healthy participants with concurrent pharmacokinetic (PK) sampling from blood plasma, urine, and cerebrospinal fluid. The overall study design is outlined below:

Part 1: Single-Dose Regimen and Fasted-Fed Crossover. For the single-dose regimen, approximately 40 healthy male or female participants will be enrolled in 1 of 5 single-dose cohorts (designated as S1 through S5, respectively) in an ascending fashion. Each cohort will consist of 8 participants randomized to CVN766 or placebo, whereby 6 participants will receive a single oral dose of CVN766 suspension, and 2 participants will receive a matching placebo suspension under overnight fasted conditions. Participants will remain fasted for 4 hours post-dose. Consumption of water is permitted as desired except for 1 hour before and after administration of Study Drug. Sentinel dosing (1 participant to receive CVN766 and 1 participant to receive placebo) will be used in each cohort to ensure adequate safety and tolerability evaluation prior to administering CVN766 or placebo to the remainder of participants within the cohort. After blinded review by the Safety Review Group (SRG) of 24-hours, post-dose safety and tolerability data from the sentinel group, the remaining 6 participants of each cohort may be dosed provided that the adverse event (AE) profile in the first 2 participants is considered acceptable. To accommodate the lumbar puncture in the S3 fasted cohort, after the sentinel group, the remaining 6 participants dosing may be staggered every two days. The planned dose levels will be 5, 15, 45, 125, and 250 mg CVN766. The SRG will review all available blinded safety, tolerability, clinical laboratory results (minimally including samples collected from participants through 72-hours post-dose), and PK data after each cohort and before subsequent dose escalation. Each following dose level may be higher, lower, or remain the same as the preceding cohort, dependent on the recommendation of the SRG.

Additional cohort(s) may be added if deemed necessary by the SRG to fully characterize the safety and tolerability of CVN766. For example, if the maximum tolerated dose (MTD) is not reached with cohort S5, additional cohorts with higher dose levels may be considered. Such additional cohorts will follow the same schedule of events as cohorts S1 through S5. Additional/alternative PK timepoints may be implemented if the SRG determines this is necessary to fully characterize the PK profile of CVN766.

To assess the effect of food on CVN766 bioavailability in suspension formulation, single-dose administration will be repeated in a single cohort (S3) after ingestion of a standardized high-fat, high-calorie meal according to FDA Guidance for Industry (Food-effect bioavailability and fed bioequivalence studies, Dec 2002). Once the safety of the S3 cohort dose level has been assessed, the S3 cohort participants will return to the clinic (no sooner than 14 days after their prior dose, or at least 4 half-lives, has lapsed based on preliminary PK data, whichever is longer). They will receive the same dose as before, administered after ingesting a standardized breakfast. Participants will finish the entire content of their breakfast within 25 minutes and will receive CVN766 30 minutes (± 5 minutes) after beginning the meal. Sentinel dosing will not be required for participants returning to the clinic for the fed regimen. If the CVN766 PK parameters in the fasted S3 cohort reveal poor absorption with inconclusive results, the fed cohort will be deferred until a higher dose level.

Participants for all cohorts will be admitted to the study unit 1 day prior to dosing and remain in the unit for safety and PK assessments. On Day 1, participants will undergo safety monitoring and PK sampling from blood plasma through 72 hours post-dose and, for cohort S3 (fasted) only, from CSF via lumbar puncture at 3 hours post-dose. The total confinement period will be 4 nights, unless extended at the discretion of the Investigator, e.g., for monitoring and/or management of AEs. Follow-up assessments will occur on approximately Days 8 and 14 and +21 and +28 for cohort S3.

Part 2: Multiple-Dose Regimen. For the multiple-dose regimen, approximately 24 healthy male and female participants age 18 to 50 years old will be enrolled in 1 of the 3 multiple-dose cohorts (designated as M1 through M3, respectively) in an ascending fashion. The dose levels planned to be studied in the multiple-dose regimen are 45, 125, and 250 mg CVN766 for multiple-dose cohorts M1 through M3, respectively. Each multiple-dose cohort will consist of 8 participants randomized to CVN766 or placebo, whereby 6 participants will receive a daily oral dose of CVN766, and 2 participants will receive a matching placebo for 7 days. Dosing will be administered in the fasting state; this can be changed by the SRG if exposure is found to be higher in the fed state. The planned dosing duration for the multiple-dose cohorts is 7 days. However, the duration may be increased to ≤14 days at the discretion of the SRG if preliminary PK data suggests steady-state will not be achieved within 6 days of daily dosing. For each dose on intensive PK sampling days (first and last days of dosing, e.g., Days 1 and 7), participants will remain fasted for 4 hours post-dose. On other dosing days (Days 2-6), participants will remain fasted for 1-hour post-dose. Consumption of water is permitted as desired except for 1 hour before and after administration of Study Drug. Unlike the single-dose regimen, sentinel dosing within cohorts is not required in the multiple-dose regimen.

Initiation of the multiple-dose regimen will only occur after a full blinded review of all safety, tolerability, and clinical laboratory results for the fasting drug administration to single-dose Cohort S3 (minimally including samples collected through Day 4) and available PK data. For each multiple-dose cohort after the first, the actual choice of dose level may be modified by the SRG after the available blinded safety, tolerability, clinical laboratory results, and PK data in the preceding multiple-dose and corresponding single-dose cohorts (i.e., multiple-dose Cohort M2 will not initiate until the data review for multiple-dose Cohort M1 and single-dose cohort S4 is complete). Each subsequent dose level may be higher, lower, or remain the same as the preceding.

Additional multiple-dose cohort(s) may be added if deemed necessary by the SRG to fully characterize the safety and tolerability of CVN766. Such additional cohorts will follow the same schedule of events as for prior multiple-dose cohorts. Additional/alternative PK timepoints may be implemented if the SRG determines this is necessary to fully characterize the PK profile of CVN766.

Participants for all multiple-dose cohorts will be admitted to the study unit 1 day prior to dosing and remain in the unit for the duration of the dosing period and for at least 48 hours after the last dose for safety and PK assessments before discharge. On treatment Days 1 and 7, participants will undergo safety monitoring and PK sampling from blood plasma through 48 hours post-dose and, in cohort M1 only, from urine through 24 hours post-dose. In cohorts M1 and M2, on treatment Day 7 (or last day of dosing, if extended beyond Day 7), participants will undergo additional PK sampling from CSF via lumbar puncture at 3 hours post-dose. If necessary to resolve questions arising from prior cohorts' data, participants in cohort M3 may also, at SRG discretion, undergo PK sampling from CSF via lumbar puncture, with the choice of day (e.g., Day 1 or Day 7) and sampling time to be decided by SRG. Participants in MAD cohorts may be asked to return to the clinic for an additional PK sample 3 days after the last dose (e.g., Day 10) depending on emerging PK data, (i.e., t½). The total confinement period will be 9 nights unless extended for additional dosing days or management of AEs. Follow-up assessments will occur approximately 7 and 14 days after the final dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant eligibility is determined according to the following criteria prior to entry into the study:

  1. In the investigator's opinion, the participant can understand and sign the Informed Consent Form and comply with all protocol requirements.
  2. The participant is a healthy male or female adult who is 18 to 55 years of age, inclusive at the time of ICF.
  3. Participant weighs at least 45 kg (99 lbs) and has a BMI between 18.0 and 32.0 kg/m2, inclusive at Screening.
  4. A male participant who is nonsterilized* and sexually active with a female partner of childbearing potential* agrees to use adequate contraception* from signing the ICF throughout the study and for 12 weeks after the last dose.

     *Definitions and acceptable methods of contraception are defined in Section 9.1.9 Contraception and Pregnancy Avoidance Procedure, and reporting responsibilities are defined in Section 9.1.10 Pregnancy.
  5. A female participant of childbearing potential who complies with contraception requirements* or a female with no childbearing potential, defined as the participant has been surgically sterilized (hysterectomy, bilateral oophorectomy, or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 years and FSH>40 IU/L).

Exclusion Criteria: Any participant who meets any of the following criteria will not qualify for entry into the study:

1. Participant has received any investigational compound within 30 days prior to the first dose of study medication or within 5 half-lives, whichever is greater.
2. Participant is a study site employee or an immediate family member of a study site employee.
3. Participant has evidence of CS neurologic, cardiovascular, pulmonary, hepatic, hematopoietic disease, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, serious allergy, full-body allergic skin rash (including hives), psychiatric disorder, or other abnormality that may impact the ability of the participant to participate or potentially confound the study results.
4. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking CVN766 or a similar drug in the same class or that might interfere with the conduct of the study.
5. Participant has a known hypersensitivity to any component of the formulation of CVN766.
6. Participant has a positive urine result for drugs of abuse at Screening or Inpatient Check-in (Day -1).
7. Participant has a history of drug abuse or a history of alcohol abuse (more than 14 units/week) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Participant has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table as listed in Table 3: Excluded Medications and Dietary Products.
9. Male participants who do not agree to all the following rules: when sexually active with a female partner(s) of childbearing potential during the study, and for 12 weeks after the last dose of study drug: a) must use an acceptable method of birth control (condom or surgical sterilization) and b) refrain from sexual activity with female partners who do not use an acceptable method of birth control. Barrier contraception (condom) must be used by all-male participants who were not surgically sterilized at least 90 days prior to screening. Male participants must also agree to refrain from sperm donation during the study and until 12 weeks after the last dose of study drug.
10. Female participants who are pregnant or breastfeeding or plan to become pregnant or donate ova during the study or 30 days after the last dose of the study drug. Women of childbearing potential must agree to practice an acceptable method of birth control (e.g., oral or parenteral contraceptives, intrauterine device, barrier, abstinence).

    *Definitions and acceptable methods of contraception are defined in Section 9.1.9, Contraception and Pregnancy Avoidance Procedure, and reporting responsibilities are defined in Section 9.1.10, Pregnancy.
11. Participant has previously had a seizure or convulsion (lifetime, with the exception of febrile seizures), including absence seizure.
12. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, any surgical intervention known to impact absorption [e.g., bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [i.e., more than once per week] occurrence of heartburn).
13. Participant has a history of cancer or other malignancy, except for basal cell carcinoma or squamous cell carcinoma that has been in remission for at least 3 years prior to Day 1.
14. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or a human immunodeficiency virus infection at Screening.
15. Participant who regularly use nicotine-containing products (including but not limited to cigarettes, electronic cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum). Casual user may participate but must agree to refrain from the time of Screening through the duration of the study or a positive urine cotinine test at Inpatient Check-in (Day 1).
16. Participant has poor peripheral venous access (defined as more than three failed attempts to cannulate).
17. Participant has donated or lost 450 mL or more of their blood volume (including plasmapheresis) or had a transfusion of any blood product within 45 days prior to Day 1.
18. Participant has an abnormal (CS) ECG at Screening or Inpatient Check-in (Day -1). Entry of any participant with an abnormal (NCS) ECG must be approved and documented by signature by the Investigator or medically qualified sub-investigator.
19. Participant has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 40 to 90 mm Hg for diastolic, confirmed with repeat per PI discretion, at the Screening Visit or Inpatient Check-in (Day -1).
20. Participant has a resting heart rate outside the range of 40 to 100 bpm, confirmed with repeat per PI discretion, at the Screening Visit or Inpatient Check-in (Day -1).
21. Participant has a QT interval with Fridericia's correction method (QTcF) >450 ms (males) or >470 ms (females) or PR outside the range of 120 to 220 ms, confirmed with one repeat testing at the Screening Visit or Inpatient Check-in (Day -1) Visit.
22. Participant has abnormal Screening or Inpatient Check-in (Day -1) laboratory values that suggest a CS underlying disease or participant with the following lab abnormalities: ALT and/or AST >1.5 the ULN, confirmed with one repeat testing.
23. Participant has a risk of suicide according to the investigator's clinical judgment or has made a suicide attempt in the previous 2 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio Vitolo, MD, Study Chair — Cerevance
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 1 site in Australia.
Pre-assignment Details: This was a randomized, double-blind, placebo-controlled, safety, tolerability and pharmacokinetic study of escalating single ascending dose (SAD) and multiple ascending doses (MAD) of CVN766 in Healthy participants. Participants were randomized 6:1 (SAD) and 6:2 (MAD) to CVN766 or placebo.
Groups:
- SAD CVN766 5 Milligrams (mg): Participants were randomized to receive a single dose of 1 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- SAD CVN766 15 mg: Participants were randomized to receive a single dose of 15 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- SAD CVN766 45 mg: Participants were randomized to receive a single dose of 45 mg CVN766 oral suspension under overnight fasted and fed condition. Participants remained fasted for 4 hours post dose.
- SAD CVN766 125 mg: Participants were randomized to receive a single dose of 125 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- SAD CVN766 250 mg: Participants were randomized to receive a single dose of 250 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- SAD Placebo: Participants were randomized to receive a single dose of matching placebo oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- MAD CVN766 45 mg: Participants were randomized to receive a daily dose of 45 mg CVN766 oral suspension in fasting or fed state for 7 days, which was determined by the Safety Review Group (SRG).
- MAD CVN766 125 mg: Participants were randomized to receive a daily dose of 125 mg CVN766 oral suspension in fasting or fed state for 7 days, which was determined by the SRG.
- MAD CVN766 250 mg: Participants were randomized to receive a daily dose of 250 mg CVN766 oral suspension in fasting or fed state for 7 days, which was determined by the SRG.
- MAD Placebo: Participants were randomized to receive a daily dose of matching placebo oral suspension in fasting or fed state for 7 days, which was determined by the SRG.
Period: SAD Cohort 1: 5 mg (14 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 6 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SAD Cohort 2: 15 mg (14 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SAD Cohort 3: 45 mg (14 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SAD Cohort 4: 125 mg (14 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SAD Cohort 5: 250 mg (14 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD Cohort 1: 45 mg (21 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD Cohort 2: 125 mg (21 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD Cohort 1: 250 mg (21 Days)
Arm/Group | SAD CVN766 5 Milligrams (mg) | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all participants who were enrolled and received study drug.
Groups:
- SAD CVN766 5 mg: Participants were randomized to receive a single dose of 1 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- SAD CVN766 45 mg: Participants were randomized to receive a single dose of 45 mg CVN766 oral suspension under overnight fasted condition. Participants remained fasted for 4 hours post dose.
- Total: Total of all reporting groups
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (5.3) | 30.8 (7.4) | 29.8 (6.4) | 26.8 (6.5) | 26.8 (3.8) | 31.9 (13.3) | 37.2 (7.5) | 27.5 (7.6) | 31.5 (8.1) | 26.8 (4.8) | 30.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 1 | 3 | 5 | 1 | 3 | 1 | 2 | 19
  Male | 3 | 6 | 6 | 5 | 3 | 5 | 5 | 3 | 5 | 4 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 6
  Not Hispanic or Latino | 4 | 5 | 6 | 5 | 5 | 10 | 5 | 4 | 6 | 5 | 55
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 4 | 3 | 4 | 5 | 3 | 6 | 4 | 4 | 4 | 4 | 41
  Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 2 | 1 | 2 | 4 | 2 | 2 | 2 | 2 | 19
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Indigenous Australian or Torres Strait Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other, Mixed White Indigenous Australian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting at Least One Treatment-emergent Adverse Event (TEAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as any AE with onset occurring within 30 days (onset date - last date of dose + 1 ≤30) after study drug administration. Percentage of participants reporting at least one TEAE has been presented.
Time Frame: Up to Day 14
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6
Percentage of participants | 50.0 | 33.3 | 83.3 | 16.7 | 66.7 | 50.0 | 66.7 | 33.3 | 66.7 | 33.3

2. Primary Outcome: Percentage of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Blood and urine samples were collected for the analysis of laboratory parameters including clinical chemistry, hematology, and urinalysis. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 14
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings including heart rate and measured PR, QRS, QT, QT interval with Fridericia's correction method (QTcF) and QT interval with Bazett's correction method (QTcB) intervals. 12-lead ECG recordings were obtained after the participants have rested for at least 5 minutes in supine position. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 14
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Clinically Significant Abnormal Vital Signs
Description: Vital signs including blood pressure (systolic and diastolic blood pressure), pulse rate, body temperature, respiratory rate and weight were measured after the participants have rested for at least 5 minutes in supine position. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Up to Day 14
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Maximum Plasma Concentration (Cmax) (Tmax) After Single Dose Administration of CVN766
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of CVN766. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Predose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48, and 72 hours postdose at Day 1
Population: PK Population: included all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 0.9165 [0.500 to 1.100] | 1.0000 [0.500 to 1.500] | 1.0000 [0.500 to 1.500] | 1.5000 [1.050 to 2.000] | 1.5000 [1.033 to 3.000]

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 (AUC24) After Single Dose Administration of CVN766
Description: Blood samples were collected at indicated time points for PK analysis of CVN766. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Predose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16 and 24 hours postdose at Day 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours*nanograms per milliliter | 319.904 (25.0) | 2155.879 (31.6) | 4001.523 (37.0) | 10990.192 (72.1) | 15607.247 (36.1)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC [0-infinity]) After Single Dose Administration of CVN766
Description: as for outcome 6
Time Frame: as for outcome 5
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours*nanograms per milliliter | 322.066 (25.7) | 2414.049 (43.4) | 4260.722 (37.2) | 13527.110 (98.9) | 19573.857 (39.4)

8. Secondary Outcome: Terminal Elimination Half-life (t1/2z) After Single Dose Administration of CVN766
Description: as for outcome 6
Time Frame: as for outcome 5
Population: PK Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 2.9625 (0.92895) | 7.3485 (4.57313) | 5.7745 (2.11356) | 11.4565 (10.57028) | 8.6156 (1.75924)

9. Secondary Outcome: Maximum Observed Trough Concentrations After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: At Days 1, 2, 3, 4, 5 and 6
Population: PK Population. Only those participants with data available at specified time points have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 5 | 6 | 6
Nanograms per milliliter
  Day 1 | 32.443 (94.0) | 208.061 (60.4) | 605.924 (68.1)
  Day 2 | 47.839 (90.2) | 278.564 (75.0) | 856.904 (75.1)
  Day 3 | 65.131 (65.0) | 298.945 (74.2) | 1002.607 (98.8)
  Day 4 | 61.883 (59.3) | 325.191 (76.0) | 1058.768 (108.5)
  Day 5 | 75.024 (55.5) | 330.735 (85.3) | 1075.797 (96.7)
  Day 6 | 81.352 (76.5) | 359.249 (83.3) | 1068.025 (82.9)

10. Secondary Outcome: Cmax After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: Predose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, and 24 (Day 2 predose) hours postdose at Day 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
Nanograms per milliliter | 534.420 (19.8) | 1309.959 (30.6) | 2398.089 (38.6)

11. Secondary Outcome: AUC From Time 0 to the End of Dosing Interval (AUCtau) After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: Predose (within 15 minutes prior to dosing) and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36, 48, and 72 a hours postdose at Day 7
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours*nanograms per milliliter | 5523.759 (39.3) | 18712.219 (45.8) | 42303.478 (49.5)

12. Secondary Outcome: T1/2z After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: as for outcome 11
Population: PK Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 7.7710 (3.20745) | 10.9721 (6.76714) | 12.1702 (4.47362)

13. Secondary Outcome: Accumulation Ratio (Rac) of Cmax After Repeat Dose Administration of CVN766
Description: Blood samples were collected at indicated time points for PK analysis of CVN766. PK parameters were analyzed using standard non-compartmental analysis. Rac (Cmax) was calculated as steady state Cmax at Day 7 divided by Cmax Day 1.
Time Frame: as for outcome 11
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 1.390 (13.7) | 1.528 (41.7) | 1.588 (33.7)

14. Secondary Outcome: Rac of AUC After Repeat Dose Administration of CVN766
Description: Blood samples were collected at indicated time points for PK analysis of CVN766. PK parameters were analyzed using standard non-compartmental analysis. Rac (AUC) was calculated as steady state AUC at Day 7 divided by AUC Day 1
Time Frame: as for outcome 11
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 1.627 (25.6) | 1.517 (49.3) | 1.771 (28.8)

15. Secondary Outcome: Time to Reach Steady State of CVN766 Concentration in the Dosing Interval
Description: Blood samples were collected at indicated time points for PK analysis of time to reach steady state of CVN766. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: as for outcome 11
Population: PK Population. Only those participants with data available at specified time points have been presented.
Measure: Median (Full Range); unit: hours
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Tmax, ss | 1.2750 [0.500 to 2.017] | 2.0000 [1.500 to 2.000] | 1.7415 [1.000 to 2.000]
  Tmin, ss: number analyzed (Participants) | 5 | 4 | 2
  Tmin, ss | 24.0000 [24.000 to 24.000] | 24.0000 [16.000 to 24.000] | 20.0165 [16.033 to 24.000]
  Tlast, ss | 42.0000 [16.100 to 48.083] | 48.0335 [48.000 to 73.967] | 73.2915 [48.000 to 77.767]

16. Secondary Outcome: Steady State Cmax After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: as for outcome 11
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 6 | 6 | 6
Nanograms per milliliter | 742.582 (14.8) | 2001.021 (32.9) | 3807.481 (33.2)

17. Secondary Outcome: Steady State Minimum Observed Plasma Concentration (Cmin) After Repeat Dose Administration of CVN766
Description: as for outcome 6
Time Frame: as for outcome 11
Population: PK Population. Only those participants with data available at specified time points have been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg
Number analyzed (Participants) | 5 | 6 | 6
Nanograms per milliliter | 77.760 (74.5) | 315.991 (89.7) | 1042.811 (79.0)

18. Secondary Outcome: Ratio of the CVN766 Concentration in Cerebrospinal Fluid (CSF) Versus the Plasma Concentration After Single Ascending Dose of CVN766 45 mg
Description: The CSF samples were collected at indicated time point for PK analysis of CVN766. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: At 3 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Unitless
Arm/Group | SAD CVN766 45 mg
Number analyzed (Participants) | 6
Unitless | 11.558 (31.7)

19. Secondary Outcome: Ratio of the CVN766 Concentration in CSF vs the Plasma Concentration After Repeated Dose Administration of CVN766
Description: as for outcome 18
Time Frame: At 3 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Unitless
Arm/Group | MAD CVN766 45 mg
Number analyzed (Participants) | 6
Unitless | 13.083 (25.9)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 14
Description: Safety Analysis Population: included all participants who were enrolled and received study drug.
Arm/Group | SAD CVN766 5 mg | SAD CVN766 15 mg | SAD CVN766 45 mg | SAD CVN766 125 mg | SAD CVN766 250 mg | SAD Placebo | MAD CVN766 45 mg | MAD CVN766 125 mg | MAD CVN766 250 mg | MAD Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 5/6 | 1/6 | 4/6 | 5/10 | 4/6 | 2/6 | 4/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAD CVN766 5 mg (N=6) | SAD CVN766 15 mg (N=6) | SAD CVN766 45 mg (N=6) | SAD CVN766 125 mg (N=6) | SAD CVN766 250 mg (N=6) | SAD Placebo (N=10) | MAD CVN766 45 mg (N=6) | MAD CVN766 125 mg (N=6) | MAD CVN766 250 mg (N=6) | MAD Placebo (N=6)
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Vascular access site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep talking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05105243/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT05105243/SAP_001.pdf